CLINICAL TRIAL: NCT06067308
Title: Predictive Accuracy of YEARS Score in Diagnosis of Pulmonary Embolism
Brief Title: YEARS Score vs CTPA in Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hussien Fayiad, Clinical Professor, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSC 265
Record Dates: First submitted 2023-09-15; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- to assess the sensitivity and accuracy of YEARS score in the diagnosis of PE. (Experimental): 50 patients with suspected PE were evaluated in Chest Department at faculty of medicine, Kasr Al-Ainy Hospital. At the beginning, clinical evaluation using YEARS score was done; subsequently for definitive diagnosis, computed tomography pulmonary angiography was performed in all cases as a reference method.
  Interventions: Diagnostic Test: Performance of CTPA

INTERVENTIONS:
Diagnostic Test: Performance of CTPA — Exposure to CT scan and injection of IV contrast

SUMMARY:
The investigators' aim in this study is to assess the sensitivity and accuracy of YEARS algorithm in the diagnosis of PE.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a relatively common acute cardiovascular disorder with high early mortality rates that, despite advances in diagnosis and treatment over the past 30 years, have not changed significantly. Due to pulmonary bed obstruction, PE can result in acute right ventricular (RV) failure. Because most patients ultimately die within the first hours of presentation, early diagnosis is of paramount importance.

The incidence of PE is estimated to be approximately 60 to 70 per 100,000, and that of venous thrombosis approximately 124 per 100,000 of the general population.

Because of its diagnostic accuracy and wide availability, multidetector row computed tomography pulmonary angiography (CTPA) is the imaging test of choice to confirm acute pulmonary embolism in most patients. Increasing use of CTPA with diminishing prevalence of pulmonary embolism to even less than 10% has led to overdiagnosis of mostly subsegmental pulmonary embolism and unnecessary risks of radiation exposure and contrast medium induced nephropathy.

To avoid these problems, validated diagnostic algorithms for suspected acute pulmonary embolism, using sequential testing, have been introduced. In these algorithms, a normal D-dimer test result in patients with low probability safely excludes pulmonary embolism.

YEARS scoring system is an algorithm to predict diagnosis of pulmonary embolism according to clinical signs and D-dimer. The aim of this study is to test predictive accuracy, sensitivity and specificity of YEARS score compared to CTPA in the diagnosis of PE as CTPA is an invasive procedure, expensive and not readily available in many settings, thus, finding an alternative easier method that can diagnose PE may help save the time and resources.

ELIGIBILITY:
Inclusion Criteria:

* Any patient more than 18 years old presenting to the emergency room with symptoms of clinically suspected pulmonary embolism such as:

  * Sudden onset of dyspnea, sudden deterioration of existing dyspnea, sudden onset of pleuritic chest pain without another apparent cause.
  * Any other symptoms like hemoptysis, syncope or unilateral leg pain.

Exclusion Criteria:

* Pregnancy

  * Allergy to intra-venous contrast agents
  * Renal insufficiency (creatinine clearance < 30 mL/min).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
YEARS score vs CTPA in diagnosis of PE | One year
  In patients with no YEARS items and a D-dimer concentration less than 1000 ng/mL, pulmonary embolism was considered excluded and further testing was withheld. In patients with one or more YEARS items and a D-dimer concentration less than 500 ng/mL, pulmonary embolism was also considered excluded and further testing was withheld. All other patients i.e., either with no YEARS item and a D-dimer concentration of 1000 ng/mL or more, or with one or more items and a concentration of 500 ng/mL or more were referred for CTPA to show or exclude the diagnosis of pulmonary embolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Almeida NA, de Sousa JT, Bachion MM, Silveira Nde A. [The use of respiration and relaxation techniques for pain and anxiety relief in the parturition process]. Rev Lat Am Enfermagem. 2005 Jan-Feb;13(1):52-8. doi: 10.1590/s0104-11692005000100009. Epub 2005 Mar 3. Portuguese. PMID 15761580